CLINICAL TRIAL: NCT06730776
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Dyspareunia: a Randomized Controlled Trial
Brief Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Dyspareunia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa gamal abdelrahman ahmed, Master student at Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005373
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Dyspareunia (Female)
Keywords: dyspareunia,
MeSH Terms: conditions — Dyspareunia | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (group A) (Active Comparator): It will include 19 women with dyspareunia. They will receive only topical medication (lidocaine ointment applied as required for symptoms and 30 minutes before sexual activity)
  Interventions: Other: Topical medication
- Study group (group B) (Experimental): It will include 19 women with dyspareunia. They will receive Acu-TENS (30 minutes per session, once per week for 10 weeks), topical medication(lidocaine ointment applied as required for symptoms and 30 minutes before sexual activity)
  Interventions: Other: Topical medication; Other: Transcutaneous electrical acupoint stimulation

INTERVENTIONS:
Other: Topical medication — It will be given to all participants in both groups (A&B). The most commonly prescribed topical medication is lidocaine ointment 5% (Xylocaine jelly 2% or ointment 5%; AstraZeneca Pharmaceuticals LP, Wilmington, DE), applied as required for symptoms and for 30 minutes before sexual activity.
Other: Transcutaneous electrical acupoint stimulation — This procedure will be applied for group B only. Before starting the first treatment session, each patient will be instructed briefly about the nature of the treatment to gain the patient's confidence and cooperation. This procedure will be performed by using TENS device on acupoints as the following: The participating woman will be placed in a relaxed comfortable supine position with her back well supported. The surface of the treated skin and the electrodes will be cleaned with alcohol wipe. The TENS protocol consists of a 30-minute weekly. session for 10 weeks of biphasic pulses with modulation 0/10-50 Hz of frequency and 300/100/3000 microseconds of pulse duration (s). The intensity parameter will be adapted individually according to each woman's perception, and modulated so that it is applied without discomfort, ranging between 10 and 100 mA (pulsing sensation) (Dionisi and Senatori ,2011)
  Arms: Study group (group B)

SUMMARY:
Transcutaneous electrical acupoint stimulation (TEAS)was proven to stimulate the secretion of endogenous opioid peptides which are partial substitutes for the exogenous opioids stimulated by drugs in the central nervous system and can thus relieve pain. Till now there is no previous study that investigates the effect of TEAS on dyspareunia. This study will determine the effect of transcutaneous acupoint stimulation on dyspareunia.

Patients will be divided randomly into two groups equal in number: The control group will receive only topical medication. The study group will receive Acu-TENS and topical medication.

DETAILED DESCRIPTION:
Patients will be divided randomly into two groups equal in number:

Control group (Group A): It will include 19 women with dyspareunia. They will receive only topical medication (lidocaine ointment applied as required for symptoms and 30 minutes before sexual activity).

Study group (GroupB): It will include 19 women with dyspareunia. They will receive Acu-TENS (30 minutes per session, once per week for 10 weeks), and topical medication (lidocaine ointment applied as required for symptoms and 30 minutes before sexual activity). All females will be given a full explanation of the study protocol and a consent form will be signed by each female before participating in the study

ELIGIBILITY:
* Inclusion Criteria:

  * Women complain of secondary dyspareunia, diagnosed and referred by the gynecologist.
  * Multiparous women.
  * Their ages will range from 25-35 years.
  * Their body BMI will be less than 35 kg/m².
  * Their pain level on the VAS will be ≥ 4.
  * All the women were negative for vaginal infections caused by viruses, bacteria or fungi.
* Exclusion Criteria:

  * Pregnancy
  * Malignancy.
  * The presence of an intrauterine device, vaginal infection, or skin/mucous lesions.
  * Diabetes mellitus.
  * Dermatological abnormalities on the skin at acupuncture point.
  * Severe uncontrolled cardiac patients or implanted cardiac rhythm devices.
  * Dyspareunia with endometriosis.
  * Fearing from electricity.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain intensity | Ten weeks
  Visual analogue scale (VAS) will be used to measure pain intensity for each female in both groups (A&B). Each female will be asked to mark the point on the scale that represents her pain level.
Assessment of dyspareunia | 10 Weeks
  Marinoff Dyspareunia Scale will be used to evaluate vaginal and vulvar symptoms and pain related to sexual intercourse for both groups (A& B) before and after the end of the treatment (10 weeks).

SECONDARY OUTCOMES:
Assessment of sexual function | Ten weeks
  The female sexual function index will be used to evaluate sexual function including (desire, arousal, lubrication, satisfaction, and orgasm) for all women with dyspareunia in both groups (A& B) before and after the end of the treatment.
Assessment of quality of life | Ten weeks
  Sexual quality of life-female (SQOL-F) questionnaire will be used to evaluate quality of life for all women with dyspareunia in both groups (A&B) before and after the end of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Osman, Study Chair — Department of Women's Health, Faculty of Physical Therapy, Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No